CLINICAL TRIAL: NCT01519596
Title: Minimizing Physical Function Decline in Older Adults Receiving Chemotherapy
Brief Title: Symptom-Adapted Physical Activity Intervention in Minimizing Physical Function Decline in Older Patients With Acute Myeloid Leukemia Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00019467; NCI-2012-00003 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97711 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-01-20; First posted 2012-01-27 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Counseling; Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (physical activity) (Experimental): Patients participate in an orientation session introducing the exercise program and protocol, reviewing fundamental principles, and demonstrating each activity. Patients also receive educational materials to facilitate orientation and adherence. Patients are offered 20-50 minute standard, intermediate, and/or low intensity physical activity sessions 5 days a week for 4 weeks. Patients also receive lifestyle-related counseling for 20-30 minutes once weekly.
  Interventions: Procedure: quality-of-life assessment; Other: counseling intervention; Behavioral: exercise intervention; Other: educational intervention
- Arm II (usual care) (Active Comparator): Patients undergo usual care for 4 weeks.
  Interventions: Procedure: quality-of-life assessment; Procedure: standard follow-up care

INTERVENTIONS:
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: counseling intervention — Receive lifestyle-related counseling
  Other Names: counseling and communications studies
  Arms: Arm I (physical activity)
Behavioral: exercise intervention — Undergo physical activity intervention
  Arms: Arm I (physical activity)
Other: educational intervention — Receive educational materials
  Other Names: intervention, educational
  Arms: Arm I (physical activity)
Procedure: standard follow-up care — Undergo usual care
  Arms: Arm II (usual care)

SUMMARY:
This is a randomized clinical trial that studies symptom-adapted physical activity intervention in minimizing physical function decline in older patients with acute myeloid leukemia (AML) undergoing chemotherapy. Physical activity may help decrease functional impairment and improve the quality of life in patients with AML undergoing chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of conducting a symptom-adapted, randomized behavioral intervention designed to improve physical function in older adults receiving chemotherapy for AML.

II. To estimate the effect size of the physical activity intervention on change in an objective measure of physical function, SPPB (short physical performance battery).

SECONDARY OBJECTIVES:

I. To estimate the effects of the physical activity intervention on self-reported physical function, health-related quality of life, and symptoms (depression, distress, fatigue).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients participate in an orientation session introducing the exercise program and protocol, reviewing fundamental principles, and demonstrating each activity. Patients also receive educational materials to facilitate orientation and adherence. Patients are offered 20-50 minute standard, intermediate, and/or low intensity physical activity sessions 5 days a week for 4 weeks. Patients also receive lifestyle-related counseling for 20-30 minutes once weekly.

ARM II: Patients undergo usual care for 4 weeks.

After completion of study treatment, patients are followed up every two weeks for two months and then monthly until week 24.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML with pathologic confirmation by World Health Organization (WHO) criteria
* Planned induction chemotherapy
* Absence of active medical problems that preclude participation in exercise (including, but not limited to: bleeding, acute thrombosis, ischemia, hemodynamic instability, uncontrolled pain)
* Patient must be ambulatory or able to walk with a cane
* Patients must have limited cognitive deficits (< 3 incorrect responses on the Pfeiffer Mental Status Scale)
* Adequate English skills to understand and complete questionnaires
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Presence of active medical conditions precluding participation to exercise (e.g., ischemia, bleeding, thrombosis, uncontrolled pain, hemodynamic instability)
* Inability to ambulate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-03-05 (Actual); Study Completion 2017-02-05 (Actual)

PRIMARY OUTCOMES:
Feasibility, in terms of participation rates and barriers to recruitment and retention | Approximately 4 weeks
  Number of exercise sessions completed, dropout rates, completion rates of the physical function measures, and completion rates of questionnaires will be recorded. Adherence will be defined as completion of at least 60% of the offered sessions.
Magnitude and trajectory of changes in objective physical function | Approximately 4 weeks
  Characterized using mixed model analysis of variance (ANOVA) with an appropriate error structure to account for the correlated nature of the data.

SECONDARY OUTCOMES:
Self-reported physical function using the SPPB, PAT-D, MAT-sf, grip strength, and lower extremity strength | Approximately 4 weeks
Self-reported quality of life | Approximately 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Klepin HD, Tooze JA, Rejeski WJ, Mihalko S, Pardee TS, Ellis L, Howard D, Demark-Wahnefried W, Powell BL, Kritchevsky S. Pilot study of an inpatient physical activity intervention for older adults treated intensively for acute myeloid leukemia. Blood Adv. 2025 Oct 28;9(20):5152-5163. doi: 10.1182/bloodadvances.2025016260. PMID 40737540